CLINICAL TRIAL: NCT07023003
Title: Postpartum Evaluation of Antihypertensives for Control of Hypertension: A Randomized Controlled Equivalence Study
Brief Title: Postpartum Evaluation of Nifedipine and Enalapril for Hypertension
Acronym: PEACE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nebraska Methodist Health System (Other)
Collaborators: Methodist Hospital Foundation (Unknown)
Responsible Party: Principal Investigator, Todd Lovgren, Principal Investigator, Nebraska Methodist Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 1551
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Hypertension in Pregnancy
Keywords: Hypertension; Postpartum; Enalapril; Nifedipine; Readmission
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension | interventions — Enalapril; Enalaprilat; Nifedipine

STUDY DESIGN:
Intervention Model Description: Open Label Randomized Controlled Equivalence Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nifedipine XR (Active Comparator): Patients will be randomized to receive nifedipine 30mg XR BID. Any additional changes in treatment will be at the discretion of their provider.
  Interventions: Drug: Nifedipine 30mg XL BID
- Enalapril 10mg QD (Experimental): Patients will be administered 10mg enalapril daily. Any additional intervention or changes in management of their hypertension will be at the discretion of their primary provider.
  Interventions: Drug: Enalapril 10mg QD

INTERVENTIONS:
Drug: Enalapril 10mg QD — Enalapril 10mg PO QD will be given to manage postpartum hypertension. Duration of treatment to be dictated by primary provider.
  Other Names: vasotec; enalaprilat; epaned
  Arms: Enalapril 10mg QD
Drug: Nifedipine 30mg XL BID — Nifedipine 30mg XL BID will be given to manage postpartum hypertension. Duration of treatment to be dictated by primary provider.
  Other Names: adalat; procardia
  Arms: Nifedipine XR

SUMMARY:
This is an open label, randomized controlled trial designed to compare nifedipine and enalapril in the management of postpartum hypertension. This is an equivalence study- meaning it is not expected one medication is better than the other. Nifedipine has been shown to be better than another common blood pressure medicine, labetalol, for postpartum hypertension but enalapril which is also used worldwide to manage blood pressure postpartum, has not yet been evaluated or compared to nifedipine.

Investigators will identify and offer enrollment to women who are admitted for delivery with documented hypertension- participants with either chronic hypertension or pregnancy related hypertension will be included. Our hypothesis is both medications are safe and effective in managing blood pressure and preventing readmission for hypertensive complications during the postpartum period so evaluating the rate of readmission is the primary goal of the study.

The only intervention of the trial will be to assign which medication the participant starts taking. Any decisions after that point- stopping medication, changing doses, additional medications, discharge from the hospital, etc, will all be at the discretion of the participant's primary provider.

ELIGIBILITY:
Inclusion Criteria:

1. admitted for delivery by cesarean or vaginal delivery
2. 24 weeks gestation or greater
3. Pregnancy related hypertension(HTN) or chronic hypertension. Pregnancy related hypertension will be defined during the study as either a systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg on two occasions at least 4 hours apart. This definition is consistent with the ACOG definition for pregnancy related HTN in patients without CHTN.

Exclusion Criteria:

1. Absolute contraindication to either nifedipine or enalapril Relative contraindications will be reviewed with PI.
2. Persistent HR <60 or >110
3. Native language other than English

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Hospital Readmission | Within 6 weeks of delivery
  Number of participants meeting criteria for hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Lovgren, MD, Principal Investigator — Nebraska Methodist Health System
Locations (1):
- Methodist Women's Hospital, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for data sharing will be reviewed on a case by case basis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of the study and for up to 10 years after completion assuming continued access to data is available.
Access Criteria: Access will be provided on a case by case basis. If shared, an encrypted and deidentified spreadsheet with non-identifying data will be provided.